CLINICAL TRIAL: NCT03384316
Title: Multi-Targeted Recombinant Ad5 (CEA/MUC1/Brachyury) Based Immunotherapy Vaccine Regimen in People With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julius Strauss, M.D., National Cancer Institute, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180032; 18-C-0032
Record Dates: First submitted 2017-12-23; First posted 2017-12-27 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Neoplasms; Prostate Cancer; Lung Cancer; Breast Cancer; Colon Cancer
Keywords: Combination Vaccine; Adenoviral; ETBX-011; ETBX-061; ETBX-051
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Adenoviridae Infections | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Arm 1-Dose De-Escalation (Experimental): Dose De-Escalation
  Interventions: Biological: ETBX-051; adenoviral brachyury vaccine; Biological: ETBX-061; adenoviral Mucin-1 (MUC1) vaccine; Biological: ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine
- 2/Arm 2 - Dose Expansion (Experimental): Dose Expansion
  Interventions: Biological: ETBX-051; adenoviral brachyury vaccine; Biological: ETBX-061; adenoviral Mucin-1 (MUC1) vaccine; Biological: ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine

INTERVENTIONS:
Biological: ETBX-051; adenoviral brachyury vaccine — immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Biological: ETBX-061; adenoviral Mucin-1 (MUC1) vaccine — immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Biological: ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine — immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year

SUMMARY:
Background:

ETBX-011, ETBX-061, and ETBX-051 are cancer vaccines. Their goal is to teach the immune system to target and kill cancer cells. The vaccines target 3 proteins found in many types of cancer. Researchers think targeting all 3 proteins in unison will have the best results.

Objective:

To test the safety of combining ETBX-011, ETBX-061, and ETBX-051 and their effects on the immune system.

Eligibility:

People ages 18 and older with advanced cancer that has not responded to standard therapies

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Scan: They will lie in a machine that takes pictures of the body.

Participants will receive the 3 vaccines through 3 shots under the skin every 3 weeks for 3 doses, then every 8 weeks for up to 1 year. They will have blood and urine tests at each vaccine visit. They will have scans and other measurements of their tumor after 9 weeks and then at their vaccine visits every 8 weeks.

Participants will keep a diary of symptoms at the injection site.

Participants will have a visit 90 days after their final treatment. This will include a physical exam and blood and urine tests. If they have any ongoing side effects, they will be followed until these end or are not changing.

After this visit, they will be called every 3 months for the first year, every 6 months for the next 2 years, then every 12 months for another 2 years to see how they are doing.

Participants will have the option to enroll in a long-term follow-up study.

...

DETAILED DESCRIPTION:
Background:

* The overall goal of the current project is to expand our immunotherapeutic approach for the treatment of advanced cancer employing a multi-targeted approach.
* Therapeutic cancer vaccines targeting overexpressed proteins offer a potential method to activate T cells against tumors.
* A novel adenovirus based vaccine targeting three (3) human tumor associated antigens (TAA), carcinoembryonic antigen (CEA), mucin-1 (MUC1), and brachyury, respectively has demonstrated anti-tumor cytolytic T cell responses in pre-clinical animal models of cancer.

Objectives:

-To determine the overall safety and recommended phase 2 dose of a combination of three immunotherapeutic vaccines (ETBX-011/ETBX-061/ETBX-051), when administered subcutaneously (SC) to subjects with advanced solid tumors

Eligibility:

* Subjects age 18 and older with cytologically or histologically confirmed locally advanced or metastatic solid tumor malignancy who have completed or had disease progression on at least one prior line of disease-appropriate therapy or who are not candidates for therapy of proven efficacy for their disease.
* Subjects may have measurable or non-measurable but evaluable disease. Subjects with surgically resected metastatic disease at high risk of relapse are also eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Adequate organ and bone marrow function
* Subjects with active autoimmune diseases requiring systemic treatment and subjects requiring systemic steroids (except for physiologic doses for steroid replacement) are not allowed

Design:

* This is a Phase I trial in subjects with advanced cancer. A combination of three therapeutic vaccines (ETBX-011, ETBX-51, EBX-61) using the same modified Adenovirus vector backbone, separately encoding three well-studied tumor-associated antigens will be assessed. The vaccine will be tested at a single dose level, and a dose de-escalation design (if required). The dose level of each vaccine tested will be 5x1011 VP. This dose has been found in prior phase 1 testing of Ad5 [E1-, E2b-]-CEA(6D) (ETBX-011) to be well tolerated (with no dose-limiting toxicities (DLTs) or related Serious adverse events (SAEs), and optimal for induction of immune responses. Each of the three vaccines will be administered subcutaneously (SC) at separate injection sites (proximal limb, preferably the thigh), every 3 weeks for 3 doses, then bi-monthly (every 8 week) boosts for up to a year.
* Up to six patients will be enrolled at Dose Level 1. If less than or equal to l of 6 patients experience a DLT, initiation of the dose expansion phase will occur. If greater than or equal to 2 of 6 experience DLT at Dose Level 1, then dose de-escalation will occur. Up to six patients will be enrolled at the lower dose level Dose Level -1 (1x10^11 VP). If less than or equal to 1 of 6 patients experience a DLT, then the maximum tolerated (MTD) will be declared at this dose, and initiation of the dose expansion phase will occur. If greater than or equal to 2 of 6 experience DLT at Dose Level -1, then a protocol amendment may be written to evaluate a further dose de-escalation.
* A dose expansion phase of study will be enrolled after the MTD of the combination vaccine has been determined. An additional 4 subjects will be enrolled in the dose expansion component of the trial, for a total of 10 subjects at the MTD.
* The ETBX-011, ETBX-51 and ETBX-61 vaccines will be administered SC every 3 weeks for 3 doses, and then bi monthly boosts for up to a year. Evaluations including immunological assessments will be carried out at baseline, on days of vaccination, and after the last vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years (male and female).
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board (IRB)'s guidelines.
* Subjects with cytologically or histologically confirmed locally advanced or metastatic solid tumor malignancy.
* Subjects must have completed or had disease progression on at least one prior line of disease-appropriate therapy or not be candidates for therapy of proven efficacy for their disease.
* Subjects may have measurable or non-measurable but evaluable. Subjects with surgically resected locally advanced or metastatic disease at high risk of relapse are also eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1.
* Subjects who have received prior carcinoembryonic antigen (CEA), mucin-1 (MUC1), and/or Brachyury-targeted immunotherapy (vaccine) are eligible for this trial if this treatment was discontinued at least 4 weeks prior to enrollment.
* Resolution of clinically significant side effects of prior chemotherapy, radiotherapy, immunotherapy or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria in Adverse Events (CTCAE) Grade less than or equal to 1 or grade less than or equal to 2 for neuropathy.

  * Adequate hematologic function at screening, as follows:
  * Absolute neutrophil count (ANC) >= 1 x 10^9/L
  * Hemoglobin >= 9 g/dL
  * Platelets >= 75,000/mcL.
* Adequate renal and hepatic function at screening, as follows:

  * Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) >= 40 mL/min (if using the Cockcroft-Gault formula below):

    * Female CrCl = ((140 - age in years) x weight in kg x 0.85) / (72 x serum creatinine in mg/dL)
    * Male CrCl = ((140 - age in years) x weight in kg x 1.00)/ 1.00) / (72 x serum creatinine in mg/dL)
  * Bilirubin less than or equal to 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 x ULN, unless liver metastases are present, then values must be less than or equal to 3 x ULN)
* The effects of the combination ETBX-011, ETBX-051, ETBX-061 vaccine regimen on the developing human fetus are unknown. For this reason, female subjects of childbearing potential defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or who is not postmenopausal (menopause being defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes) and male patients who are not surgically sterile (vasectomy etc.), must agree to use acceptable contraceptive methods for the duration of the study and for one month after the last vaccination. Acceptable forms of contraception include oral contraceptives, intrauterine device, condom or vaginal diaphragm plus spermicidal (gel/foam/cream/vaginal suppository), or total abstinence.
* Ability to attend required study visits and return for adequate follow up, as required by this protocol.

EXCLUSION CRITERIA:

* Pregnant and nursing women. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with combination ETBX-011, ETBX-051, ETBX-061, breastfeeding should be discontinued if the mother is treated with combination ETBX-011, ETBX-051, ETBX-061. These potential risks may also apply to other agents used in this study.
* There should be a minimum of 4 weeks from any prior investigational drug, chemotherapy, immunotherapy, with the exception of hormonal therapy for prostate and breast cancers, human epidermal growth factor receptor 2 (HER2-) directed therapy for HER2+ breast or stomach cancer (3+ immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH+), drugs targeting epidermal growth factor receptor (EGFR), anaplastic large-cell lymphoma kinase (ALK) or ROS1 in EGFR,ALK, ROS1-mutated lung cancer, respectively, or standard maintenance therapies for any solid tumor under the condition that subjects are on these therapies for at least two months before start of trial treatment.
* There should also be a minimum of 4 weeks from any prior radiotherapy except for palliative bone directed therapy.
* Known active brain or central nervous system metastasis (less than 1 month out from definitive radiotherapy or surgery), or seizures requiring anticonvulsant treatment, or clinically significant cerebrovascular accident or transient ischemic attack (<3 months).
* Subjects with active autoimmune disease requiring systemic immunosuppressive treatment within the past 4 weeks such as but not restricted to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. A history of autoimmune disease which is not active nor has required recent systemic immunosuppressive therapy (< 4 weeks prior to enrollment) is not reason for exclusion.
* Subjects with serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, or other illness considered by the Investigator as high risk for investigational drug treatment.
* Subjects with clinically significant heart disease, such as congestive heart failure (class II, III, or IV defined by the New York Heart Association functional classification), history of unstable or poorly controlled angina, or history (< 1 year) of ventricular arrhythmia.
* Subjects with a medical or psychological impediment that would impair the ability of the subject to receive therapy per protocol or impact ability to comply with the protocol or protocol-required visits and procedures.
* History of second malignancy within 3 years prior to enrollment except for the following: adequately treated non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer or other localized malignancy after discussion with the medical monitor.
* Presence of a known active acute or chronic infection, including human immunodeficiency virus (HIV, as determined by enzyme-linked immunosorbent assay (ELISA) and confirmed by western blot) and hepatitis B and hepatitis C virus (HBV/HCV, as determined by hepatitis B surface antigen (HBsAg) and hepatitis C serology).
* Subjects on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (less than or equal to the equivalent of prednisone 10 mg/day) or other immunosuppressives such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 2 weeks prior to enrollment for recent short course use (less than or equal to 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (> 14 days). In addition, the use of corticosteroids as premedication for contrast-enhanced studies is allowed prior to enrollment and on study.
* Subjects with known allergy or hypersensitivity to any component of the investigational product will be excluded.
* Subjects with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
* Subjects vaccinated with a live (attenuated) vaccine (e.g., FluMist(R)) or a killed (inactivated)/subunit vaccine (e.g., PNEUMOVAX(R), Fluzone(R)) within 28 days or 14 days, respectively, of the first planned dose of ETBX vaccine.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Y Strauss, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balint JP, Gabitzsch ES, Rice A, Latchman Y, Xu Y, Messerschmidt GL, Chaudhry A, Morse MA, Jones FR. Extended evaluation of a phase 1/2 trial on dosing, safety, immunogenicity, and overall survival after immunizations with an advanced-generation Ad5 [E1-, E2b-]-CEA(6D) vaccine in late-stage colorectal cancer. Cancer Immunol Immunother. 2015 Aug;64(8):977-87. doi: 10.1007/s00262-015-1706-4. Epub 2015 May 9. PMID 25956394
- [Background] Morse MA, Chaudhry A, Gabitzsch ES, Hobeika AC, Osada T, Clay TM, Amalfitano A, Burnett BK, Devi GR, Hsu DS, Xu Y, Balcaitis S, Dua R, Nguyen S, Balint JP Jr, Jones FR, Lyerly HK. Novel adenoviral vector induces T-cell responses despite anti-adenoviral neutralizing antibodies in colorectal cancer patients. Cancer Immunol Immunother. 2013 Aug;62(8):1293-301. doi: 10.1007/s00262-013-1400-3. Epub 2013 Apr 30. PMID 23624851
- [Background] Gabitzsch ES, Tsang KY, Palena C, David JM, Fantini M, Kwilas A, Rice AE, Latchman Y, Hodge JW, Gulley JL, Madan RA, Heery CR, Balint JP Jr, Jones FR, Schlom J. The generation and analyses of a novel combination of recombinant adenovirus vaccines targeting three tumor antigens as an immunotherapeutic. Oncotarget. 2015 Oct 13;6(31):31344-59. doi: 10.18632/oncotarget.5181. PMID 26374823
- [Result] Gatti-Mays ME, Redman JM, Donahue RN, Palena C, Madan RA, Karzai F, Bilusic M, Sater HA, Marte JL, Cordes LM, McMahon S, Steinberg SM, Orpia A, Burmeister A, Schlom J, Gulley JL, Strauss J. A Phase I Trial Using a Multitargeted Recombinant Adenovirus 5 (CEA/MUC1/Brachyury)-Based Immunotherapy Vaccine Regimen in Patients with Advanced Cancer. Oncologist. 2020 Jun;25(6):479-e899. doi: 10.1634/theoncologist.2019-0608. Epub 2019 Oct 8. PMID 31594913
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0032.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP): Up to 6 patients will be enrolled on Dose Level 1. If ≤1 of 6 patients experience a dose limiting toxicity, initiation of the Dose Expansion phase will occur.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
  ETBX-061; adenoviral Mucin-1 (MUC1) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
  ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
- Expansion Cohort - 5 x 10^11 Viral Particles (VP): ≤1 of 6 patients experienced a dose limiting toxicity on Dose Level 1, thus subjects were enrolled in a Dose Expansion phase.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-061; adenoviral Mucin -1 (MUC1) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Period: Overall Study
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Screen failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Expansion Cohort - 5 x 10^11 Viral Particles (VP): ≤1 of 6 patients experienced a dose limiting toxicity on Dose Level 1, thus subjects were enrolled in a Dose Expansion phase.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-061; adenoviral Mucin-1 (MUC1) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (8.1) | 48.6 (12.9) | 49.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11
Number of Participants with Adenovirus 5-Neutralizing Antibodies [Count of Participants; unit: Participants] — Population: Serum for antibody analysis was only available for 5/6 participants in the Dose Level 1 Cohort, and 3/5 participants in the Expansion Cohort.
  Participants
    number analyzed (Participants) | 5 | 3 | 8
    (all) | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 16 months and 6 days.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP): Up to 6 patients will be enrolled on Dose Level 1. If ≤1 of 6 patients experience a dose limiting toxicity, initiation of the Dose Expansion phase will occur.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-061; adenoviral Mucin -1 (MUC1) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants | 6 | 4

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: RP2D is defined as ≤ 1 of 6 of the initial 6 subjects who experience a dose limiting toxicity (DLT), than this dose level will be defined as the RP2D. A DLT is defined as any Grade 3 or greater toxicity that is possibly related to the vaccine and as defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 with the exception of transient (≤ 24 hours) Grade 3 flu-like symptoms or fever, which is controlled with medical management (≤ 24 hours) Grade 3 fatigue, skin reactions or rash, headache, nausea, emesis that resolves to Grade ≤ 1 or asymptomatic grade 3 amylase/lipase elevation.
Time Frame: RP2D was based upon evaluation of DLTs. Participants were followed for DLTs from the first dose of vaccine for 3 weeks.
Population: RP2D was determined in Dose Level 1 cohort.
Measure: Number; unit: billion viral particles per indiv. vacc.
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6
billion viral particles per indiv. vacc. | 500

3. Secondary Outcome: Number of Participants Who Achieve an Objective Confirmed Complete or Partial Response Assessed by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Objective response is determined by participants whose tumors shrunk after therapy assessed by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately 3.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants
  Confirmed Complete Response | 0 | 0
  Partial Response | 0 | 0

4. Secondary Outcome: Number of Patients With Disease Control (Confirmed Response or Stable Disease (SD)) Lasting for at Least 6 Months
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for Partial Response (PR) nor sufficient increase to qualify for Progressive Disease (taking as reference the smallest sum diameters while on study).
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants | 1 | 1

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The amount of time a subject survives without disease progression after treatment. Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum diameters while on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of 5 mm. (Note: the appearance of one or more lesions is also considered progression).
Time Frame: up to 12 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
weeks | 10 [3 to 22] | 9 [6 to 30]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the amount of time a subject survives after therapy assessed from the date of first treatment to the date of death (any cause).
Time Frame: up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
months | 9.5 [2.0 to NA] — There are insufficient events after the median to calculate the upper bound. It is 'not estimable'. | 9.5 [5.0 to NA] — There are insufficient events after the median to calculate the upper bound. It is 'not estimable'.

7. Other Pre Specified Outcome: Number of Participants With a Positive Mucin-1 (MUC-1) Specific T-Cells Immune Response
Description: Peripheral blood mononuclear cells (PBMC) were analyzed by flow cytometry to evaluate anti-tumor response induced by vaccine injection.
Time Frame: up to week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants | 3 | 3

8. Other Pre Specified Outcome: Number of Participants With a Positive Carcinoembryonic Antigen (CEA) Specific T-Cells Immune Response
Description: as for outcome 7
Time Frame: up to week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants | 2 | 2

9. Other Pre Specified Outcome: Number of Participants With a Positive Brachyury Specific T-Cells Immune Response
Description: as for outcome 7
Time Frame: up to week 6
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP): Up to 6 patients will be enrolled on Dose Level 1. If ≤1 of 6 patients experience a dose limiting toxicity, initiation of the Dose Expansion phase will occur.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
  ETBX-061; adenoviral MUC1 vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
  ETBX-011; adenoviral CEA vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Participants | 1 | 2

10. Other Pre Specified Outcome: Number of Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as any Grade 3 or greater toxicity that is possibly related to the vaccine and as defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 with the exception of transient (≤ 24 hours) Grade 3 flu-like symptoms or fever, which is controlled with medical management (≤ 24 hours) Grade 3 fatigue, skin reactions or rash, headache, nausea, emesis that resolves to Grade ≤ 1 or asymptomatic grade 3 amylase/lipase elevation.
Time Frame: From the date of the first dose of vaccine, approximately 3 weeks.
Measure: Number; unit: Toxicities
Groups:
- Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP): Up to 6 patients will be enrolled on Dose Level 1. If ≤1 of 6 patients experience a dose limiting toxicity, initiation of the Dose Expansion phase will occur.
  ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously ETBX-051; adenoviral brachyury vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-061; adenoviral Mucin -1 (MUC1) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year ETBX-011; adenoviral Carcinoembryonic antigen (CEA) vaccine: immunotherapeutic vaccine administered subcutaneously every 3 weeks for 3 doses, and then every 8 weeks for up to a year
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
Number analyzed (Participants) | 6 | 4
Toxicities | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 16 months and 6 days.
Arm/Group | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) | Expansion Cohort - 5 x 10^11 Viral Particles (VP)
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) (N=6) | Expansion Cohort - 5 x 10^11 Viral Particles (VP) (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Infections and Infestations - Other, Gram-negative bacteremia, 40 degree C fever (Infections and infestations) | 1 (1) | 0 (0)
Death, NOS (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Cohort - 5 x 10^11 Viral Particles (VP) (N=6) | Expansion Cohort - 5 x 10^11 Viral Particles (VP) (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2)
Flu like symptoms (General disorders) | 5 (5) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 6 (6) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 5 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03384316/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03384316/Prot_SAP_001.pdf